CLINICAL TRIAL: NCT05291364
Title: The Effectiveness of Adding Dexmedetomidine to Alcohol in Splanchnic Nerve Neurolysis for the Treatment of Intra-Abdominal Cancer Pain.
Brief Title: Dexmedetomidine in Splanchnic Nerve Neurolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, haidy salah mansour, associate professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 673-8/2020
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Dexmedetomidine
Keywords: Splanchnic Nerve Neurolysis; Chronic cancer Pain
MeSH Terms: interventions — Dexmedetomidine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): injection of ethanol and lidocaine with dexmedetomidine
  Interventions: Drug: Group 1
- Group 2 (Active Comparator): injection of ethanol and lidocaine Without dexmedetomidine
  Interventions: Drug: Group 2

INTERVENTIONS:
Drug: Group 1 — Is formed of 20 patients had splanchnic plexus block with 4.5 ml ethanol 96% + 1.5 ml of lidocaine 10 mg/ml + 2 μg/kg dexmedetomidine diluted in 0.9% sterile saline (total volume 12 ml) on each side
  Other Names: dexmedetomidine
  Arms: Group 1
Drug: Group 2 — Is formed of 20 patients had splanchnic plexus block with 4.5 ml ethanol 96% + 1.5 ml of lidocaine 10 mg/ml diluted in 0.9% sterile saline (total volume 12 ml) on each side.
  Other Names: ethanol
  Arms: Group 2

SUMMARY:
Malignancy related abdominal and pelvic pain can be debilitating and affects survival as well as quality of life. Pain from cancer and its treatments can result in anxiety, depression, fear, anger, helplessness, and hopelessness, and those with both pain and depression have an amplification of disability and poor quality of life Pancreatic and other upper abdominal organ malignancies can produce intense visceral pain syndromes that are frequently treated with splanchnic nerve neurolysis (SNN) or celiac plexus neurolysis (CPN). Dexmedetomidine is a selective alpha two adreno-receptor agonist. It provides dose-dependent sedation, analgesia, sympatholysis, and anxiolysis without relevant respiratory depression. Dexmedetomidine is used as adjuvant to LA drugs in peripheral nerve block, brachial plexus block and intrathecal anesthesia with satisfactory results. The aim of this study is to evaluate effect of addition of dexmedetomidine as an adjuvant to alcohol and local anesthetics for chemical neurolysis to control pain in patients with intra-abdominal malignancy.

DETAILED DESCRIPTION:
Patients fasted for 6 hours prior to the procedure, and a 20 G intravenous cannula was placed. Before the procedure, 500 mL of physiological saline was administered intravenously. The patient was positioned in the prone position on the surgical table with the chest supported using a pillow, to reverse the thoracolumbar lordosis and to increase the distance between the superior iliac spine and the chest cage. The patient was monitored using electrocardiography, non-invasive blood pressure measurements, and pulse oximetry in accordance with the standards proposed by the American Association of Anesthesiologists. On arrival at the operating room, electrocardiogram, pulse oximetry, and non-invasive arterial blood pressure were applied and vital signs were obtained.

Twenty-two Gauge spinal needle introduced at 11th intercostal space 6 cm from midline and advanced to touch the anterolateral aspect of T11. Again, with AP and lateral views the placement of the needles was confirmed using contrast dye under fluoroscopy.

Splanchnic nerve blockade will be performed by using (4.5 ml ethanol 96% + 1.5 ml of lidocaine 10 mg/ml) administered bilaterally (a total volume of 12 ml) with addition of 2 μg/kg dexmedetomidine patients in group (1).

The procedure lasted 30 minutes, and the recovery period lasted 10 minutes since conscious sedation was used. After the procedure, patients were kept under medical observation for 4 to 6 hours to monitor possible hemodynamic complications.

Parameters assessed:

1. Hemodynamic parameters: Heart rate, respiratory rate and oxygen saturation were recorded before and immediately after the blockade and follow up on time intervals over 2 weeks after the blockade.
2. Analgesic requirements: First time to require additional analgesics
3. Visual Analogue Scale: The Visual Analogue Scale score (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'.The score of pain intensity was determined by patients providing a mark between 0-10 cm with score from 0-4 cm mild pain. 5- 7 cm moderated and 8-10 severe pain
4. Incidence of complications: In the form of hemodynamic instability, constitutional symptoms as (nausea, vomiting and diarrhea)

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed to have abdominal malignancy aged 25 to 70 years old
* Fully conscious
* Patient has no hematological disease or coagulation abnormality.
* Patient has no history of mental illness
* Patient with persistent and moderate to severe abdominal pain visual analogue scale score > 4.

Exclusion Criteria:

* Patient refusal of the procedure
* Extremes of age
* Patients with psychiatric disorders
* Patient diagnosed to have any coagulation defect or bleeding tendency
* Patients with cardiopulmonary significant condition
* Skin infection or wounds at site of proposed needle insertion site

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 2 weeks
  Visual Analogue Scale which measure the pain intensity . It determined by patients providing a mark between 0-10 cm with score from 0-4 cm mild pain. 5- 7 cm moderated and 8-10 severe pain. it was recorded prior to injection and after injection by 6,12,24,72 hours and after one and two weeks

SECONDARY OUTCOMES:
the time of analgesic requirement | 2 weeks
  measure the time with hours passes after the injection to require additional analgesics as tramadol

CONTACTS AND LOCATIONS:
Overall Officials: Haidy S Mansour, Study Director — Associate professor
Locations (1):
- Minya University, Minya, Egypt